CLINICAL TRIAL: NCT06646718
Title: Effect Of Closed Kinetic Chain On Hip Stability In Spastic Cerebral Palsy Post Selective Dorsal Rhizotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Shaza Salah Eldin Ahmed Mostafa Elabd, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KFSIRB200-171
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy; Selective Dorsal Rhizotomy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: * The study will include children (age 5-14years) post selective dorsal rhizotomy.
  * Children meeting the inclusion criteria will be randomly assigned to one of two groups:
    * Experimental Group: children in this group will receive closed kinetic chain.
    * Control Group: Patients in this group will receive Traditional physical therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ❖ Experimental Group: group A (Experimental): Group A (study group): will include 33 children after selective dorsal rhizotomy surgery from both gender will be selected from the Outpatient Clinic. Able to attend physical therapy (PT) treatment at least three a week before and during this study. who will receive closed kinetic chain.
  Interventions: Procedure: Close kinetic chain exercise group
- ❖ Control Group:Group B (Other): ●Group B (control group): will include 33 children who will receive Traditional physiotherapy. will include 33 children after selective dorsal rhizotomy surgery from both gender
  Interventions: Procedure: Traditional physical therapy.

INTERVENTIONS:
Procedure: Close kinetic chain exercise group — ●Close kinetic chain exercise group: group A will receive forward step-ups, lateral step-ups, squats, sit-to-stand, and stoop-and-recover exercises. session will be initiated with a 10 min warm-up period, including stretching of the major muscles and muscle groups, then 40 min different exercises and terminated with a 10 min cool-down period in the form of aerobic exercises.
  Other Names: Experimental group intervention
  Arms: ❖ Experimental Group: group A
Procedure: Traditional physical therapy. — ●Traditional physiotherapy: group B will receive stretching for the lower extremity muscles, namely hip flexors and adductors, hamstrings, and calf muscles; and strengthening exercises for core muscles, hip extensors, flexors and abductors, internal and external rotators of the hip, flexors and extensors of the knee, ankle dorsi flexors, kneeling exercises, and standing and gait training
  Other Names: Control group intervention
  Arms: ❖ Control Group:Group B

SUMMARY:
Purpose of the study:

To evaluate the effect of closed kinetic chain on hip stability after selective dorsal rhizotomy on spastic cerebral palsy.

DETAILED DESCRIPTION:
* This is a prospective randomized controlled clinical trial, conducted at Kafr El sheikh Hospital.
* Sixty-six children of both genders.
* The study will include children (age 5-14years) post selective dorsal rhizotomy.
* Children meeting the inclusion criteria will be randomly assigned to one of two groups:

  * Experimental Group: children in this group will receive closed kinetic chain.
  * Control Group: Patients in this group will receive Traditional physical therapy.
* Randomization will be achieved using computer-generated random numbers to ensure an equal distribution of patients between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients will be aged from 5 to 14 years

  2- will be included both genders post selective dorsal rhizotomy.

  3- The GMFCS level I-II spastic diplegia, able to stand up from a chair independently and maintain standing for more than 5 seconds without falling.

  4- Had not received any strength training program in the past 3 months before the study.

  5- Able to attend physical therapy (PT) treatment at least three a week before and during this study.

Exclusion Criteria:

* 1-have perceptual, cognitive, visual and auditory disorder.

  2- botulinum toxin injection to the lower extremities within 6 Months.

  3- Medical conditions that prevented children from participating in the exercises.

  4- Previous lower extremity surgery, such as prior hamstring muscle Lengthening. 5- Existence of any orthopedic condition or any static hip, knee or ankle deformities.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-10-12 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Isokinetic dynamometry: | 12 weeks
  Isokinetic dynamometry testing is a device used within sports and exercise science as well as clinical testing environments that is used to evaluate joint torque. Isokinetic dynamometers are able to test the strength (torque) and power of different muscle groups.
  is a safe and reliable method accepted as the "gold standard" in the evaluation of muscle strength.
  It will be used before and after intervention to measure muscle strength
X-ray: | 12 weeks
  used to assess the alignment of the hip joint, detect any abnormalities, and determine the degree of bone deformities or hip dislocation.
  Will be used before and after intervention to determine hip angles
The Pediatric Balance Scale: | 12 weeks
  The Pediatric Balance Scale (PBS), which is a modification of Berg Balance Scale (BBS) designed for children and adolescents aged 5 to 15 years, to assess functional balance abilities. The scale is composed of 14 items that are scored on a criterion-based 0 to 4 scale. The range of scores in the PBS is 0 to 56. each activity is rated on a five-point scale (0-4) so that the maximum score is 56. Patients who score 41 or higher are considered to be a low fall risk, those who score between 21 and 40 are considered to be moderate fall risks, and those who score below 20 are considered to be high fall risks. It will be completed in 15-20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Abdelaziz Ali Sherief, Professor, Study Director — Kafr elsheikh University
Locations (1):
- Faculty of physical therapy, Kafr elsheikh University, Kafr ash Shaykh, Kafr Elsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No